CLINICAL TRIAL: NCT05521230
Title: Randomised Clinical Trial on the Short-Term Anti-plaque Effect of Cymenol Mouthwash Analysed Using Dentius Deep Plaque Software
Brief Title: Short-Term Anti-plaque Effect of Cymenol Mouthwash Analysed Using Dentius Deep Plaque Software
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Lacer S.A. (Industry)
Responsible Party: Principal Investigator, Inmaculada Tomás, Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021_CE112
Record Dates: First submitted 2022-07-25; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Healthy; Dental Plaque
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants rinsed 10 ml of placebo mouthwash for a period of 60 seconds, three times a day with an interval of 7-9 hours in between, for 4 days (period 1)
  Interventions: Drug: Placebo Mouthwash
- Cymenol (test) (Experimental): Participants applied a 10 ml rinse of 0.1% cymenol mouthwash for a period of 60 seconds, three times a day with a 7-9 hour interval in between, for 4 days (period 1) and 4 days more (period 2)
  Interventions: Drug: Cymenol mouthwash

INTERVENTIONS:
Drug: Placebo Mouthwash — Application of mouthwashes
  Arms: Placebo
Drug: Cymenol mouthwash — Application of mouthwashes
  Arms: Cymenol (test)

SUMMARY:
The objective of this project was to investigate the short-term in situ anti-plaque effect of cymenol, using the Dentius Deep Plaque software

ELIGIBILITY:
Inclusion criteria were as follows:

* Systemically healthy volunteers
* Age between 20-45 years
* Presence of minimum of 24 permanent teeth
* No evidence of gingivitis or periodontitis (CPITN= 0)
* No presence of untreated caries at the start of the study.

Exclusion criteria were as follows:

* Smoker or ex-smoker
* Presence of dentures or orthodontic appliances
* Antibiotic treatment in the last 3 months or routine use of oral antiseptics

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in the plaque area: baseline vs 4 days | Baseline, 4 days
  Change in the percentage of the tooth surface with dental plaque:baseline vs 4 days
Change in the plaque area: baseline vs 8 days | Baseline, 8 days
  Change in the percentage of the tooth surface with dental plaque: baseline vs 8 days
Change in the plaque area: 4 days vs 8 days | 4 days, 8 days
  Change in the percentage of the tooth surface with dental plaque: 4 days vs 8 days
Change in the growth rate of dental plaque area: baseline vs 4 days | Baseline, 4 days
  Change in the growth rate of dental plaque area (percentage area/hour): baseline vs 4 days
Change in the growth rate of dental plaque area: baseline vs 8 days | Baseline, 8 days
  Change in the growth rate of dental plaque area (percentage area/hour): baseline vs 8 days
Change in the growth rate of dental plaque area: 4 days vs 8 days | 4 days vs 8 days
  Change in the growth rate of dental plaque area (percentage area/hour): 4 days vs 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Tomás, Prof., Principal Investigator — University of Santiago de Compostela, Spain
Locations (1):
- University of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suarez-Rodriguez B, Regueira-Iglesias A, Blanco-Pintos T, Balsa-Castro C, Vila-Blanco N, Carreira MJ, Tomas I. Short-term anti-plaque effect of a cymenol mouthwash analysed using the DenTiUS Deep Plaque software: a randomised clinical trial. BMC Oral Health. 2023 Aug 12;23(1):560. doi: 10.1186/s12903-023-03256-9. PMID 37573292